CLINICAL TRIAL: NCT01614873
Title: Comparison of Breathing Pattern During PSV and NAVA
Brief Title: Comparison of Breathing Pattern During Neurally Adjusted Ventilatory Assist Ventilation and Pressure Support Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Collaborators: Adep Assistance (Other)
Responsible Party: Principal Investigator, Lofaso, MD-PhD, Centre d'Investigation Clinique et Technologique 805
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2012-A0030043
Record Dates: First submitted 2012-06-06; First posted 2012-06-08 (Estimated); Last update posted 2013-04-12 (Estimated); Status verified 2013-04

CONDITIONS: Respiratory System Abnormalities
Keywords: Breathing Pattern; Mechanical Ventilation; Pressure support ventilation; Neurally Adjusted Ventilatory Assist
MeSH Terms: conditions — Respiratory System Abnormalities | interventions — Critical Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pressure Support Ventilator (Active Comparator): Gold standard partial ventilator support: Pressure Support Ventilation performed with Servo-i® ventilator (MAQUET,Critical Care, Sweden).
  During pressure support the inspiratory muscles are assisted by a constant inspiratory pressure adjusted by the prescriptor and applied to the airway by either an invasive or a non invasive interface. Then the subject initiate the inspiratory effort and a constant pressure is delivered to the airway in order to assist inspiration. Three levels of pressure will be tested (5 cmH2O, 8 cmH2O and 12 cmH2O)
  Interventions: Device: Servo-i® ventilator, MAQUET,Critical Care, Sweden
- NAVA (Experimental): Spontaneous Breathing using Neurally Adjusted Ventilatory Assist with trigger adjusted on diaphragmatic electromyogram. Electrical activity of the diaphragm will be obtained through a naso-gastric tube with multiple array of electrodes placed at its distal end (Eadi catheter® , Maquet Critical Care, Sweden). During NAVA the inspiratory muscles are assisted by a pressure which is proportional to this electrical activity. Then the subject initiate the inspiratory effort and a pressure proportional to the integrated EMG activity is delivered to the airway in order to assist inspiration. The adjustment of the level of NAVA (expressed in cmH2O/microvolt) will be adjusted in order to obtain a peak pressure similar to pressure support (5 cmH2O, 8 cmH2O and 12 cmH2O)
  Interventions: Device: Servo-i® ventilator, MAQUET,Critical Care, Sweden

INTERVENTIONS:
Device: Servo-i® ventilator, MAQUET,Critical Care, Sweden — Electrical activity of the diaphragm will be obtained through a naso-gastric tube with multiple array of electrodes placed at its distal end (Eadi catheter® , Maquet Critical Care, Sweden). Subject will be ventilated with a mouthpiece interface. NAVA will be compared to Pressure Support using the same ventilator. Once the pattern of breathing will be stabilized (10 minutes) in each condition (see arm) the following parameters will be recorded during 5 minutes and compared : tidal volume, inspiratory time, expiratory time, transcutaneous CO2 pressure, diaphragmatic Emg activity, delay between the inspiratory activity initiation and positive pressure initiation, delay between the end of the inspiratory effort and the end of pressurisation.
  Other Names: PSV

SUMMARY:
Comparison of Breathing pattern during mechanical ventilation. Two modes of mechanical ventilation are compared (Pressure Support Ventilation and Neurally Adjusted Ventilatory Assist)

DETAILED DESCRIPTION:
Eligibility : healthy subject without respiratory complications in the past

Subjects will breath spontaneously without mechanical ventilation, with Pressure Support Ventilation and with Neurally Adjusted Ventilatory Assist during.

Three levels of pressurisation will be tested : 5 cmH2O, 8 cmH2O and 12 cmH2O Duration of each condition will be about 15 minutes.

Measurements will include:Flow, airway pressure, SaO2, PtCO2, diaphragmatic electromyography, chest wall motion by optoelectronic plethysmography

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Healthy Subject without any chronic disease

Exclusion Criteria:

* Absence of consent
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-05; Primary Completion 2012-05 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Comparison of breathing pattern during pressure support and Neurally Adjusted Ventilatory Assist (NAVA) | 2h

SECONDARY OUTCOMES:
Tidal volume evaluated by optoelectronic plethysmography | 2h
Electrical diaphragmatic activity recorded by mechanical ventilator | 2h

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Lofaso, MD-PhD, Principal Investigator — Hopital Raymond Poincare - Garches - France; Nicolas Terzi, MD-PhD, Principal Investigator — CHU de Caen - INSERM U1075 - France; Pascale Calabrese, PhD, Study Director — Laboratoire TIMC-IMAG - La Tronche - France; Henri Meric, Principal Investigator — EA 4497 - Hopital Raymond Poincare - Garches -France
Locations (1):
- Hopital Raymond Poincare, Garches, France

REFERENCES:
- [Derived] Meric H, Calabrese P, Pradon D, Lejaille M, Lofaso F, Terzi N. Physiological comparison of breathing patterns with neurally adjusted ventilatory assist (NAVA) and pressure-support ventilation to improve NAVA settings. Respir Physiol Neurobiol. 2014 May 1;195:11-8. doi: 10.1016/j.resp.2014.01.021. Epub 2014 Feb 5. PMID 24508509